CLINICAL TRIAL: NCT05089097
Title: Assessment of Postoperative Delirium With CAM ICU Score in Patients Treated With Serotoninergic Reuptake (SSRI) Inhibitors and Undergoing Intervention of Heart Surgery on Pump
Acronym: DeCAMS-ON
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.Cch.19.01
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Delirium
Keywords: Delirium; Postoperative; CAM-ICU Score
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhibitors of serotoninergic reuptake on: patients with a diagnosis of depressive syndrome requiring treatment with Inhibitors of serotoninergic reuptake drugs excluding neurodegenerative diseases and on treatment with antidepressants for more than three months.
  Intervention: evaluation of the presence of postoperative delirium with the CAM-ICU score upon awakening and for the following 48 hours.
  Interventions: Other: evaluation of delirium with CAM-ICU Score
- Inhibitors of serotoninergic reuptake off: patients without a diagnosis of depressive syndrome requiring treatment with Inhibitors of serotoninergic reuptake drugs excluding neurodegenerative diseases and not in treatment with antidepressants.
  Intervention: evaluation of the presence of postoperative delirium with the CAM-ICU score upon awakening and for the following 48 hours.
  Interventions: Other: evaluation of delirium with CAM-ICU Score

INTERVENTIONS:
Other: evaluation of delirium with CAM-ICU Score — the CAM-ICU score is an evaluation tool to verify the presence or absence of delirium in a subject

SUMMARY:
The study aims to observe the presence of postoperative delirium in patients undergoing elective cardiac surgery, without changing the pharmacological prescriptions of the enrolled patients and the procedures carried out by normal clinical practice.

ELIGIBILITY:
Inhibitors of serotoninergic reuptake on

Inclusion Criteria:

* patients over 18 years old
* patients undergoing elective cardiac surgery
* patients diagnosed with depressive syndrome requiring treatment with Inhibitors of serotoninergic reuptake excluding neurodegenerative diseases
* patients on antidepressant therapy for more than 3 months at the time of enrollment

Exclusion Criteria:

* absence of written informed consent to the study
* patients undergoing non-elective and emergency cardiac surgery
* patients undergoing off pump surgery
* patients with depression not on therapy
* patients with existing malignancies
* patients with acute infections in progress
* patients with previous stroke, cerebral haemorrhage with relics
* patients with acquired and congenital metabolic pathologies with CNS alterations
* Patients with acute and / or chronic renal failure according to RIFLE score (exclude only F-L-E)
* Patients with acute and / or chronic hepatic insufficiency according to Child - Pugh score <6 (but without encephalopathy);
* Patients with neurodegenerative diseases (dementias of all types both organic and vascular, parkinson's and ongoing delirium);
* Patients with previous or current drug and / or alcohol abuse
* pregnant or postpartum period patients (6 months after delivery)

Inhibitors of serotoninergic reuptake off

Inclusion Criteria:

* patients over 18 years old
* patients undergoing elective cardiac surgery
* patients without a diagnosis of depressive and psychiatric illness requiring treatment with psychoactive drugs to the exclusion of neurodegenerative diseases

Exclusion Criteria:

* absence of written informed consent to the study
* patients undergoing non-elective and emergency cardiac surgery
* patients undergoing off pump surgery
* patients with depression not on therapy
* patients with existing malignancies
* patients with acute infections in progress
* patients with previous stroke, cerebral haemorrhage with relics
* patients with acquired and congenital metabolic pathologies with CNS alterations
* Patients with acute and / or chronic renal failure according to RIFLE score (exclude only F-L-E)
* Patients with acute and / or chronic hepatic insufficiency according to Child - Pugh score <6 (but without encephalopathy);
* Patients with neurodegenerative diseases (dementias of all types both organic and vascular, parkinson's and ongoing delirium);
* Patients with previous or current drug and / or alcohol abuse
* pregnant or postpartum period patients (6 months after delivery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 18 years of age, of both sexes, undergoing elective cardiac surgery and with the presence or absence of depressive pathology in therapy with Inhibitors of serotoninergic reuptake
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Presence/absence of postoperative delirium | 4 june 2020 to 4 june 2021
  presence / absence of postoperative delirium, assessed with CAM-ICU, from awakening and for the following 48 hours

SECONDARY OUTCOMES:
Correlation with ICU-Length of Stay | 4 june 2020 to 4 june 2021
  Correlation with ICU-Length of Stay
correlation with Hospital-Length of Stay | 4 june 2020 to 4 june 2021
  correlation with Hospital-Length of Stay
Bleeding | 4 june 2020 to 4 june 2021
  measure of bleeding in ml / day
re-operated patient | 4 june 2020 to 4 june 2021
  Number of re-operated patient
mechanical ventilation in intensive care | 4 june 2020 to 4 june 2021
  number of patients who required mechanical ventilation in the ICU
mortality | 4 june 2020 to 4 june 2021
  mortality at 28 days
infections | 4 june 2020 to 4 june 2021
  number and type of infections that occurred following the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Nazionale SS Antonio e Biagio e Cesare Arrigo, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: No